CLINICAL TRIAL: NCT03556020
Title: A Randomized, Double-Blind, Parallel Group, Phase 2 Study to Assess the Safety, Tolerability, and Efficacy of Once Weekly Subcutaneous (SC) Injections of a Sustained-Release Vasoactive Intestinal Peptide (VIP) Analogue, Pemziviptadil (PB1046), in Adult Subjects With Symptomatic Pulmonary Arterial Hypertension (PAH)
Brief Title: Phase 2 Study to Assess Safety, Tolerability and Efficacy of Once Weekly SC Pemziviptadil (PB1046) in Subjects With Symptomatic PAH
Acronym: VIP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated: Study drug resupply delayed (Covid-19)
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB1046-PT-CL-0004
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — VIP-ELP fusion molecule PB1046

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose Group (Experimental): Maximally tolerated dose Drug: Pemziviptadil (PB1046), Once Weekly Subcutaneous Injection
  Interventions: Drug: Pemziviptadil (PB1046)
- Low Dose Group (Experimental): Minimally effective dose Drug: Pemziviptadil (PB1046), Once Weekly Subcutaneous Injection
  Interventions: Drug: Pemziviptadil (PB1046)

INTERVENTIONS:
Drug: Pemziviptadil (PB1046) — Pemziviptadil (PB1046), Once Weekly Subcutaneous Injection

SUMMARY:
This is a multi-center, randomized, double-blind, controlled, Phase 2 study to assess the safety, tolerability, and efficacy of pemziviptadil (PB1046) at the optimally titrated dose after 16 weeks of treatment. Subjects will be randomized in a 2:1 ratio to one of two parallel dose groups: a) high-dose group where PB1046 will be up-titrated from a 0.2 mg/kg minimally effective starting dose to a target high dose level of at least 1.2 mg/kg or higher to a maximally tolerated dose (MTD), or b) a low-dose group that will start at 0.2 mg/kg and remain at this minimally effective dose (MED) level with sham up-titration. The total treatment period will be comprised of 2 phases: 1) an initial 10 week dose titration phase in which weekly doses of PB1046 will be titrated (or sham titrated) up to a target dose level of at least 1.2 mg/kg or higher to the MTD, and 2) a maintenance of treatment phase that begins when subjects reach week 11 and continues for 6 weeks during which no further up-titration should occur.

DETAILED DESCRIPTION:
The primary safety and tolerability objectives will be assessed by investigating the incidence and severity of adverse events (AEs) as well as changes from baseline in vital signs, laboratory parameters, ECGs and their relationship to pemziviptadil (PB1046). The primary efficacy objective will be assessed by investigating the change in PVR derived from right heart catheterization (RHC). Secondary efficacy objectives will be assessed by investigating the impact of pemziviptadil (PB1046) on change from baseline in 6 minute walk distance (6MWD) test and NT-proBNP, a prognostic biomarker for PAH, in the two groups (comparing the MTD and MED groups) at the end of the treatment period. In addition, the effect of pemziviptadil (PB1046) on other cardiopulmonary hemodynamic parameters (e.g. CI, mPAP, mRAP, wedge pressure and SvO2) as measured by RHC will be assessed. Changes in BDI, HRQoL, and NYHA/WHO (New York Heart Association/World Health Organization) FC will also be assessed.

An independent Data Safety Monitoring Board (DSMB) will periodically assess safety, efficacy and biomarker data to independently assess the overall safety profile of pemziviptadil (PB1046), to help adjudicate potential dose-limiting toxicities, and to monitor the overall benefit risk profile of pemziviptadil (PB1046) during the study. The DSMB will review the safety and tolerability data after the first 10 subjects while recruitment is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with PAH, ≥18 and ≤ 79 years of age, who are symptomatic and have reduced exercise capacity due primarily to their PAH diagnosis and have been assessed by a qualified individual (i.e. physician, physician assistant, nurse practitioner) to be in NYHA/WHO functional class II or III;
* Willing and able to sign a written informed consent prior to all study-related procedures;
* Subjects with PAH belonging to one of the following subgroups of the Nice Clinical Classification of Pulmonary Hypertension Group 1: a. Idiopathic, b. Heritable, c. Drug or toxin-induced, d. Associated with connective tissue disease, HIV infection, portal hypertension, congenital heart disease (pulmonary-to-systemic shunt;
* Two 6MWD test results > 50 m and < 550 m prior to randomization with results +/- 10% of each other. Note: Up to four tests may be conducted between Screening and Randomization for eligibility purposes;
* Hemodynamic assessment of PAH demonstrating elevated mPAP and PVR as indicated below during the Screening Period: a. mean pulmonary artery pressure (mPAP) of ≥ 25 mmHg; and, b. pulmonary vascular resistance (PVR) ≥ 400 dyne•sec/cm5; and, c. pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) of ≤ 12 mmHg if PVR ≥ 400 and < 500 dynes•sec/cm5; or PCWP/LVEDP ≤ 15 mmHg if PVR ≥ 500 dynes•sec/cm5;
* Body mass index ≥ 18 kg/m2 and ≤ 40 kg/m2 at screening;
* Meet the following criteria determined by pulmonary function tests completed no more than 24 weeks prior to screening: a. Forced expiratory volume in one second (FEV1) ≥ 55% of predicted normal, b. FEV1: FVC (forced vital capacity) ratio ≥ 0.60;
* Agrees to use a medically acceptable method of contraception (both male and female patients) throughout the entire study period and continuing for 30 days after their last dose of study drug;
* Stable background medical regimen of up to 3 oral PAH therapies for at least 30 days prior to Screening and having been on PAH therapy for at least 3 months;
* If a subject has historical diagnosis (prior to screening visit) of being positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV), must be clinically stable and if on therapy, must be on stable therapy for HIV or HCV for at least 3 months; Willing and able to understand and follow instructions; return to the study unit for specified study visits; and able to participate in the study for the entire period.

Exclusion Criteria:

* Concomitant medical disorder, condition, or history, that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study;
* Concomitant medical disorder that is expected to limit the subject's life-expectancy to ≤ 1 year;
* Pregnant or lactating female subjects;
* First positive result from serology testing at visit 1 (screening labs) for HIV, HBsAg, or HCV prior to randomization;
* Participation in another investigational drug study within 30 days prior to screening or participating in a non-medication study which, in the opinion of the Investigator, would interfere with the study compliance or outcome assessments;
* Use of chronic subcutaneous prostanoid/prostacyclin therapy for PAH within 30 days prior to screening, including prostacyclin receptor agonists;
* More than mild mitral or aortic valve disease, left ventricular ejection fraction < 50%, or left ventricular regional wall motion abnormality suggestive of active coronary artery disease on documented 2D-echocardiography occurring within 12 months of Screening;
* Sustained systolic blood pressure (SBP) < 95 mmHg and/or diastolic blood pressure (DBP) < 50 mmHg (confirmed by a duplicate seated reading) on at least 3 consecutive readings (self-monitored or office) at screening and prior to dosing, or overt symptomatic hypotension;
* Sustained resting heart rate >110 beats per minute (BPM) (confirmed by duplicate assessments of office vital signs or consecutive ECG assessments) on at least 3 consecutive readings at screening and prior to dosing;
* Clinically significant renal dysfunction at the Screening Visit as measured by the estimated glomerular filtration rate (eGFR)
* Significant liver dysfunction as measured by any one of the following at screening: a. alanine aminotransferase (ALT) >3.0 times upper limit of normal (ULN) or; b. aspartate aminotransferase (AST) >3.0 times ULN or; c. serum bilirubin ≥ 1.6 mg/dL;
* Known history of substance abuse within the past 1 year that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study;
* Any major surgical procedure within 90 days prior to screening or planned surgical procedure during the study period;
* Any in-patient hospitalization (defined as greater than 23 hours) within 30 days of subject screening;
* Enrollment within the past 3 months prior to screening or plans to enroll during the study into a cardiopulmonary rehabilitation program;
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining voluntary consent or would confound the objectives of study;
* Known hypersensitivity to study drug or any of the excipients of the drug formulation;
* More than two of the following: a. BMI > 35; b. Current atrial fibrillation; c. Current Diabetes Mellitus; d. Current hypertension; e. History of clinically significant coronary artery disease in prior 3 years.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
Incidence of Clinical Laboratory Abnormalities | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
Changes in Diastolic Blood Pressure | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
Changes in Systolic Blood Pressure | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
Changes in Oral Body Temperature | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
Changes in Respiratory Rate | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
Changes in Heart Rate | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
12-Lead ECG - Incidence of clinically significant findings | 172 days - Starting up to 30 days prior to first dose and completing 28 days after last dose.
Immunogenicity | 172 days - Starting up to 30 days prior to first dose and completing 8 weeks after last dose. May be extended in the event that result does not return to baseline in time allotted.
Change in baseline in pulmonary vascular resistance (PVR) | 142 days - Pre-dose (up to 30 days prior to first dose) and post-dose 16.

SECONDARY OUTCOMES:
Change from baseline in 6MWD | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in NT-proBNP | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in cardiac index (CI) | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in mean pulmonary artery pressure (mPAP) | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in mean right atrial pressure (mRAP) | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in wedge pressure | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in mixed venous oxygen saturation (SvO2) | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in pulmonary artery compliance | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.

OTHER OUTCOMES:
Change from baseline in Borg Dyspnea Index (BDI) at the end of treatment | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change from baseline in emPHasis-10 (HRQoL) score at the end of treatment | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Change in NYHA/WHO Functional Class (FC) at the end of treatment | 142 days - Pre-dose (up to 30 days prior to first dose) and one week post-dose 16.
Incidence of clinical worsening over 16 weeks as defined by any one of the following (See description): | 142 days - Pre-dose (up to 30 days prior to first dose) and post-dose 16.
  All-cause mortality, Hospitalization due to worsening of PAH, Initiation of parenteral prostacyclin, Worsening of PAH either by >15% decrease in 6MWD or new or worsening right heart failure (RHF), or worsening of symptoms requiring escalation of PAH therapy
Time to clinical worsening with data censored at the end of treatment | 142 days - Pre-dose (up to 30 days prior to first dose) and post-dose 16.
Change from baseline in other PAH biomarkers at the end of treatment | 142 days - Pre-dose (up to 30 days prior to first dose) and post-dose 16.
Multi-dose pharmacokinetic (PK) profile of individually dose-titrated pemziviptadil (PB1046) administered once-weekly for 16 weeks - Cmax | Pre-dose (Dose 1), day 28 pre-dose, day 70 pre-dose, day 77 pre-dose, day 84 pre-dose, day 91 pre-dose, day 98 pre-dose, day 105 pre-dose, 1 and 3 hours post-dose, day 106, day 107, day 108, day 110 and day 112.
Multi-dose pharmacokinetic (PK) profile of individually dose-titrated PB1046 administered once-weekly for 16 weeks - Tmax | Pre-dose (Dose 1), day 28 pre-dose, day 70 pre-dose, day 77 pre-dose, day 84 pre-dose, day 91 pre-dose, day 98 pre-dose, day 105 pre-dose, 1 and 3 hours post-dose, day 106, day 107, day 108, day 110 and day 112.
Multi-dose pharmacokinetic (PK) profile of individually dose-titrated pemziviptadil (PB1046) administered once-weekly for 16 weeks - Ctrough | Pre-dose (Dose 1), day 28 pre-dose, day 70 pre-dose, day 77 pre-dose, day 84 pre-dose, day 91 pre-dose, day 98 pre-dose, day 105 pre-dose, 1 and 3 hours post-dose, day 106, day 107, day 108, day 110 and day 112.
Multi-dose pharmacokinetic (PK) profile of individually dose-titrated pemziviptadil (PB1046) administered once-weekly for 16 weeks - Area Under Curve(0-t) [AUC(0-t)] | Pre-dose (Dose 1), day 28 pre-dose, day 70 pre-dose, day 77 pre-dose, day 84 pre-dose, day 91 pre-dose, day 98 pre-dose, day 105 pre-dose, 1 and 3 hours post-dose, day 106, day 107, day 108, day 110 and day 112.
Multi-dose pharmacokinetic (PK) profile of individually dose-titrated pemziviptadil (PB1046) administered once-weekly for 16 weeks - AUC(0-tmax) | Pre-dose (Dose 1), day 28 pre-dose, day 70 pre-dose, day 77 pre-dose, day 84 pre-dose, day 91 pre-dose, day 98 pre-dose, day 105 pre-dose, 1 and 3 hours post-dose, day 106, day 107, day 108, day 110 and day 112.
Multi-dose pharmacokinetic (PK) profile of individually dose-titrated pemziviptadil (PB1046) administered once-weekly for 16 weeks - AUC(tmax-t) | Pre-dose (Dose 1), day 28 pre-dose, day 70 pre-dose, day 77 pre-dose, day 84 pre-dose, day 91 pre-dose, day 98 pre-dose, day 105 pre-dose, 1 and 3 hours post-dose, day 106, day 107, day 108, day 110 and day 112.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - IMC - Diagnostic & Medical Clinic, LLC, Mobile, Alabama
  - Banner University Medical Center, Tucson, Arizona
  - University of California, San Diego (UCSD), La Jolla, California
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California-Davis, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - The University Miami Health Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - The Emory Clinic, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Dept of Internal Medicine, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts University, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Linder Center for Resarch and Education at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Memorial Hermann Hospital CRU affiliated with University of Texas Health Science Center at Houston - McGovern Medical School, Houston, Texas